CLINICAL TRIAL: NCT01854450
Title: Evaluation of Asymmetrical Lateral Decubitus for Rotation of Occipitoposterior Fetal Position During Labor : EVADELA Multicentre Randomized Trial
Brief Title: Evaluation of Asymmetrical Lateral Decubitus for Rotation of Occipitoposterior Fetal Position
Acronym: EVADELA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P120902; 2012-A01578-35
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Fetal Occipitoposterior Position During the Labor
Keywords: Occipitoposterior position; Maternal posturing; Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asymmetrical Lateral Decubitus (Experimental): Women in labor are postured in pronounced lateral decubitus (side opposite to the back of the fetus), with the inferior leg in extension, and the superior leg in hyperflexion
  Interventions: Other: Asymmetrical Lateral Decubitus
- control (Other): usual obstetrical care
  Interventions: Other: control

INTERVENTIONS:
Other: Asymmetrical Lateral Decubitus — After randomization, women are postured in pronounced lateral decubitus (side opposite to the back of the fetus), with the inferior leg in extension, and the superior leg in hyperflexion, during 1 hour (minimum 30 minutes).
  Then, women are encouraged to take this posture during labor as frequently as possible if the fetus remains in occipitoposterior position
  Other Names: maternal posturing
  Arms: Asymmetrical Lateral Decubitus
Other: control — usual obstetrical care
  Arms: control

SUMMARY:
Maternal posturing is used during labor to facilitate the rotation of occipitoposterior fetal position in anterior.

Our study aims to evaluate the efficacy of asymmetrical lateral decubitus for rotation of the fetal head.

DETAILED DESCRIPTION:
The prevalence of fetal occipitoposterior position during labor is 20%. Compared to anterior positions, they are known to be at higher risk of complications (cesarean section, instrumental delivery, severe perineal laceration).

Maternal posturing is used during labor to facilitate the rotation of the fetal head in anterior position. Asymmetrical lateral decubitus is used frequently, without having ever been evaluated.

Our study aims to evaluate the efficacy of this maternal posturing, through a randomized open trial.

We hypothesized that posturing women in asymmetrical lateral decubitus allows increasing frequency of anterior fetal position after 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* women older than 18 years
* Gestational age ≥ 37SA,
* Ruptured membranes,
* single living fetus in cephalic presentation with an occipitoposterior position clinically diagnosed between 2 and 9 cm dilated and confirmed by ultrasound.
* Affiliation to a social security scheme (beneficiary or assignee)
* Signing the consent

Exclusion Criteria:

* Fetal presentation other than posterior
* Multiple pregnancy,
* Breech presentation
* History of previous cesarean section
* Fetal death in utero, termination of pregnancy
* Fetal intrauterine fetal growth restriction <5e percentile,
* Fetal malformation,
* Women younger than 18 years old,
* Women do not understand French,
* Women with psychiatric condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Fetal head position | 1 hour
  fetal head position one hour after randomization

SECONDARY OUTCOMES:
fetal head position | at diagnosis of full dilatation
  Clinical evaluation of the fetal head position at diagnosis of full cervical dilatation confirmed with ultrasound
Speed of cervical dilatation | during the first stage of labour
  Duration of labor between randomization and full dilatation
Mode of delivery and perineal complications | at delivery
  Mode of delivery (spontaneous vaginal, instrumental vaginal delivery, cesarean section) and perineal complications (episiotomy, severe perineal tears).
feasibility and acceptability of asymmetrical lateral decubitus | during and after labour
  quality of fetal heart rate monitoring during maternal posturing Evaluation of maternal satisfaction using self-administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Camille Le Ray, MD, PhD, Principal Investigator — Port-Royal Maternity Hospital
Locations (4):
- France (4):
  - Maternité du CH d'Avranches-Granville, Avranches-Granville
  - CHU côte de nacre, Caen
  - Port-Royal Maternity Hospital, Paris
  - bluets maternity Hospital, Paris

REFERENCES:
- [Background] Le Ray C, Lepleux F, De La Calle A, Guerin J, Sellam N, Dreyfus M, Chantry AA. Lateral asymmetric decubitus position for the rotation of occipito-posterior positions: multicenter randomized controlled trial EVADELA. Am J Obstet Gynecol. 2016 Oct;215(4):511.e1-7. doi: 10.1016/j.ajog.2016.05.033. Epub 2016 May 27. PMID 27242201